CLINICAL TRIAL: NCT06187129
Title: Evaluation of Nerve Ultrasound in Detecting Clinical and Subclinical Peripheral Neuropathy in Children and Adolescent With Type 1 Diabetes Mellitus
Brief Title: Evaluation of Nerve Ultrasound in Detecting Clinical and Subclinical Peripheral Neuropathy in Children and Adolescents With Type 1 Diabetes Mellitus
Status: Not yet recruiting | Type: Observational
Sponsor: Esraa Hosny Dahy (Other)
Responsible Party: Sponsor-Investigator, Esraa Hosny Dahy, assistant lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Nerve ultrasound in neuropathy
Record Dates: First submitted 2023-12-16; First posted 2024-01-02 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- diabetic children and adolescent with type 1 diabetes: nerve ultrasound and nerve conduction study
  Interventions: Device: nerve ultrasound
- healthy age matched group: nerve ultrasound
  Interventions: Device: nerve ultrasound

INTERVENTIONS:
Device: nerve ultrasound — nerve ultrasound
  Other Names: nerve conduction study

SUMMARY:
Aim of study:

To evaluate accuracy of nerve ultrasound in detecting clinical and subclinical peripheral neuropathy in children and adolescents diagnosed with type 1 diabetes melitus .

DETAILED DESCRIPTION:
Introduction Type 1 diabetes (T1D) is a chronic disease with long-term vascular complications which include nephropathy, retinopathy, neuropathy, and macrovascular disease . In childhood and adolescence, early functional and structural vascular related abnormalities may be present a few years after the onset of the disease, so In this period intensive education and treatment may prevent or delay the onset and progression of complications.

Diabetic neuropathy (DN) is an important complication in patients with diabetes since it is related to mortality, morbidity, and a decrease in the quality of life ,as it is associated with neuropathic pain, foot ulceration, and subsequently gangrene and amputation.

Typical DPN is a chronic, nerve-length-dependent, distal symmetrical sensorimotor polyneuropathy (DSPN) and is considered as the most common form among diabetic neuropathies .

DPN can be classified into subclinical and clinical stages; based on history with sensory disturbances (possible); symptoms and/or signs of nerve dysfunction (probable); symptoms and/or signs plus abnormal gold standard test (confirmed); abnormal gold standard test (subclinical).

Subclinical neuropathy is defined as asymptomatic peripheral neuropathy, which is one of the common complications of patients with diabetes mellitus (DM). There is considerable uncertainty about the prevalence of diabetic peripheral neuropathy (DPN) in pediatric populations, which is probably due to the lack of large epidemiological studies performed on pediatric patients with DM, who often show few symptoms of neurological involvement.

Evidence from western studies have suggested that a quarter of children and adolescents with type 1 diabetes have clinical or subclinical evidence of nerve injury at diagnosis , The prevalence of peripheral neuropathy in known children with T1DM is reported to be as high as 50% .

Many risk factors have been suggested for peripheral neuropathy, such as the duration of diabetes, age at onset, height, puberty, positive family history, and diabetic complications of puberty .

The effect of chronic hyperglycemia is mediated by the increase of the intracellular level of glucose and sorbitol, which eventually leads to oxidative stress and the generation of free radicals, which damage intracellular macromolecules. In addition, chronic hyperglycemia induces the formation of advanced glycation end products (AGEs), which modify the structure of myelin, leading to axonal degeneration.

Currently, the diagnosis of DPN is mainly based on characteristic symptoms and signs. Nerve conduction studies (NCS) is one of the gold standard techniques for diagnosing DPN . It evaluates the occurrence and development of DPN by detecting the ability of peripheral nerve to transmit electrical signals in patients with DN. NCS has the characteristics of being quantifiable, objective, and sensitive, but it has the following disadvantages: time-consuming, high cost, poor experience, and the need for professional doctors to operate.

Although there are no guidelines on screening subclinical diabetic neuropathy, nerve conduction study (NCS) is the most common tool used for diagnosing it.

The pattern of nerve dysfunction has varied in neurophysiological studies on pediatric populations .Some studies found that subclinical sensory affection is prevalent. And others found that subclinical motor affection more common.

High-resolution ultrasound is of growing importance as a painless method complementary to nerve conduction studies in the workup of disorders of the peripheral nervous system, especially in children and adolescents .Cross-sectional area, echogenicity, morphology of the individual nerve fascicles, thickness of the epineurium, vascularization and mobility of the nerve are the main parameters evaluated with nerve ultrasound in polyneuropathies.

High-frequency ultrasound was first used in the clinical diagnosis of DPN as a supplement to NCS. It measures the size, blood vessels, echo, and mobility of the diseased nerve to show the damage of the nerve tissue, which can effectively improve the diagnostic efficiency of DPN and reduce the missed diagnosis rate and the misdiagnosis rate . In patients with DPN, the cross sectional area (CSA) and longitudinal section of the nerve are increased, and the echogenicity of the nerve, the boundary ambiguity, and the blood flow in the nerve are also significantly increased. The mean CSA in the examined nerves was higher in moderate to severe DPN than the mild DPN .

High resolution ultrasound has unique diagnostic advantages for early or subclinical neuropathy. High-frequency ultrasound can detect subclinical involvement of peripheral nerves and abnormalities in patients with normal electrical diagnosis .

ELIGIBILITY:
Inclusion Criteria:

- 1.Children and adolescents aged 8-17 y diagnosed as type 1 DM according to American diabetes association ( ADA) (17) .

2.On multiple injection or insulin pump for at least 5 years or more. 3.Patients are free from acute complication like diabetes ketoacidosis (DKA), symptomatic hypoglycemia, or infection for at least one month before enrollment in the study.

Exclusion Criteria:

* 1.Age less than 8 years or more than 17 years. 2.Diabetes other than T1DM . 3.Patients with known neuropathy of any other cause rather than diabetes. 4.Diabetic children with thyroid dysfunction ,coelic disease or anemia.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1. Children and adolescents aged 8-17 y diagnosed as type 1 DM according to American diabetes association ( ADA) (17) .
  2. On multiple injection or insulin pump for at least 5 years or more.
  3. Patients are free from acute complication like diabetes ketoacidosis (DKA), symptomatic hypoglycemia, or infection for at least one month before enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
cross sectional area of peripheral nerves using nerve ultrasound | baseline
  To evaluate accuracy of nerve ultrasound in detecting clinical and subclinical peripheral neuropathy in children and adolescents diagnosed with type 1 diabetes melitus .

REFERENCES:
- [Background] Donaghue KC, Marcovecchio ML, Wadwa RP, Chew EY, Wong TY, Calliari LE, Zabeen B, Salem MA, Craig ME. ISPAD Clinical Practice Consensus Guidelines 2018: Microvascular and macrovascular complications in children and adolescents. Pediatr Diabetes. 2018 Oct;19 Suppl 27(Suppl 27):262-274. doi: 10.1111/pedi.12742. No abstract available. PMID 30079595
- [Background] Charles M, Soedamah-Muthu SS, Tesfaye S, Fuller JH, Arezzo JC, Chaturvedi N, Witte DR; EURODIAB Prospective Complications Study Investigators. Low peripheral nerve conduction velocities and amplitudes are strongly related to diabetic microvascular complications in type 1 diabetes: the EURODIAB Prospective Complications Study. Diabetes Care. 2010 Dec;33(12):2648-53. doi: 10.2337/dc10-0456. Epub 2010 Sep 7. PMID 20823346
- [Background] Kallinikou D, Soldatou A, Tsentidis C, Louraki M, Kanaka-Gantenbein C, Kanavakis E, Karavanaki K. Diabetic neuropathy in children and adolescents with type 1 diabetes mellitus: Diagnosis, pathogenesis, and associated genetic markers. Diabetes Metab Res Rev. 2019 Oct;35(7):e3178. doi: 10.1002/dmrr.3178. Epub 2019 Jun 6. PMID 31083769
- [Background] Dyck PJ, Albers JW, Andersen H, Arezzo JC, Biessels GJ, Bril V, Feldman EL, Litchy WJ, O'Brien PC, Russell JW; Toronto Expert Panel on Diabetic Neuropathy. Diabetic polyneuropathies: update on research definition, diagnostic criteria and estimation of severity. Diabetes Metab Res Rev. 2011 Oct;27(7):620-8. doi: 10.1002/dmrr.1226. PMID 21695763
- [Background] Tesfaye S, Boulton AJ, Dyck PJ, Freeman R, Horowitz M, Kempler P, Lauria G, Malik RA, Spallone V, Vinik A, Bernardi L, Valensi P; Toronto Diabetic Neuropathy Expert Group. Diabetic neuropathies: update on definitions, diagnostic criteria, estimation of severity, and treatments. Diabetes Care. 2010 Oct;33(10):2285-93. doi: 10.2337/dc10-1303. PMID 20876709
- [Background] Altuwaijri WA, Almutair AN, AlAlwan IA, Almahdi MJ, Almasoud SD. Subclinical Neuropathy in Children With Type I Diabetes Mellitus: Tertiary Care Centre Experience. Cureus. 2022 Aug 8;14(8):e27765. doi: 10.7759/cureus.27765. eCollection 2022 Aug. PMID 35949448
- [Background] Walter-Holiner I, Barbarini DS, Lutschg J, Blassnig-Ezeh A, Zanier U, Saely CH, Simma B. High Prevalence and Incidence of Diabetic Peripheral Neuropathy in Children and Adolescents With Type 1 Diabetes Mellitus: Results From a Five-Year Prospective Cohort Study. Pediatr Neurol. 2018 Mar;80:51-60. doi: 10.1016/j.pediatrneurol.2017.11.017. Epub 2017 Dec 13. PMID 29429781
- [Background] Yu Y. Gold Standard for Diagnosis of DPN. Front Endocrinol (Lausanne). 2021 Oct 26;12:719356. doi: 10.3389/fendo.2021.719356. eCollection 2021. PMID 34764937
- [Background] Misra UK, Kalita J, Nair PP. Diagnostic approach to peripheral neuropathy. Ann Indian Acad Neurol. 2008 Apr;11(2):89-97. doi: 10.4103/0972-2327.41875. PMID 19893645
- [Background] Karsidag S, Morali S, Sargin M, Salman S, Karsidag K, Us O. The electrophysiological findings of subclinical neuropathy in patients with recently diagnosed type 1 diabetes mellitus. Diabetes Res Clin Pract. 2005 Mar;67(3):211-9. doi: 10.1016/j.diabres.2004.07.017. PMID 15713353
- [Background] Toopchizadeh V, Shiva S, Khiabani NY, Ghergherechi R. Electrophysiologic pattern and prevalence of subclinical peripheral neuropathy in children and adolescents with type I diabetes mellitus in Iran. Saudi Med J. 2016 Mar;37(3):299-303. doi: 10.15537/smj.2016.3.13625. PMID 26905353
- [Background] Singh DP, Singh P, Sharma S, Aneja S, Seth A. Point Prevalence of Peripheral Neuropathy in Children and Adolescents with Type 1 Diabetes Mellitus. Indian J Pediatr. 2022 Mar;89(3):220-225. doi: 10.1007/s12098-021-03742-4. Epub 2021 Jun 10. PMID 34109557
- [Background] Yusuf I, Mork H, Erdlenbruch B, Schellinger PD, Philipps J. Nerve ultrasound reference values in children and adolescents: Echogenicity and influence of anthropometric factors including hand volume. J Cent Nerv Syst Dis. 2023 Aug 21;15:11795735231195778. doi: 10.1177/11795735231195778. eCollection 2023. PMID 37621670
- [Background] Pitarokoili K, Gold R, Fisse AL. Nerve ultrasound for the diagnosis and follow-up of peripheral neuropathies. Curr Opin Neurol. 2023 Oct 1;36(5):373-381. doi: 10.1097/WCO.0000000000001183. Epub 2023 Jun 23. PMID 37382111
- [Background] Hajas G, Kissova V, Tirpakova A. A 10-yr follow-up study for the detection of peripheral neuropathy in young patients with type 1 diabetes. Pediatr Diabetes. 2016 Dec;17(8):632-641. doi: 10.1111/pedi.12382. Epub 2016 Mar 29. PMID 27028140
- [Background] Chiang JL, Maahs DM, Garvey KC, Hood KK, Laffel LM, Weinzimer SA, Wolfsdorf JI, Schatz D. Type 1 Diabetes in Children and Adolescents: A Position Statement by the American Diabetes Association. Diabetes Care. 2018 Sep;41(9):2026-2044. doi: 10.2337/dci18-0023. Epub 2018 Aug 9. No abstract available. PMID 30093549
- [Background] Ryan CS, Conlee EM, Sharma R, Sorenson EJ, Boon AJ, Laughlin RS. Nerve conduction normal values for electrodiagnosis in pediatric patients. Muscle Nerve. 2019 Aug;60(2):155-160. doi: 10.1002/mus.26499. Epub 2019 May 11. PMID 31032944
- [Background] Grimm AS, Schubert C, Grimm A, Stahl JH, Kupper H, Horber V, Kegele J, Willikens S, Wittlinger J, Serna-Higuita L, Winter N, Groeschel S. Normative Observational Nerve Ultrasound Values in School-Age Children and Adolescents and Their Application to Hereditary Neuropathies. Front Neurol. 2020 Apr 28;11:303. doi: 10.3389/fneur.2020.00303. eCollection 2020. PMID 32411079